CLINICAL TRIAL: NCT05219877
Title: Comparison of the Effectiveness of Preurodynamic Single Dose of Levofloxacin With Posturodynamic Levofloxacin for Three Days on the Incidence of Urinary Tract Infections
Brief Title: Effectiveness of Preurodynamic With Posturodynamic Levofloxacin on the Incidence of UTI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Harrina Erlianti Rahadjo, Sp.U(K), PhD, Prof. dr., Sp.U(K), PhD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 341/UN2.F1/ETIK/PPM.00.02/2021
Record Dates: First submitted 2022-01-20; First posted 2022-02-02 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-02

CONDITIONS: Urinary Tract Infections
Keywords: Urodynamics; Antibiotics; Prophylaxis
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with a single-blinded randomized clinical trial design to compare the proportion of UTIs in a group of patients receiving levofloxacin 500 mg single dose one hour before urodynamic examination and patients receiving levofloxacin 500 mg once daily for three days post-urodynamic examination. To determine the sample treatment group, blocked randomization technique is used in this study.
Who Masked: Outcomes Assessor
Masking Description: This study uses a single-blinded design because the outcome assessed in this study is urinalysis which is the objective outcome. The urinalysis evaluator is blinded to the drug regimen obtained by the research subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-urodynamic Levofloxacin (Experimental): Levofloxacin 500 mg single dosage 1 hour before the urodynamic examination
  Interventions: Drug: Pre-urodynamic Levofloxacin
- Post-urodynamic Levofloxacin (Active Comparator): Levofloxacin 500 mg will be given for 3 days, once daily, post-urodynamic examination
  Interventions: Drug: Post-urodynamic Levofloxacin

INTERVENTIONS:
Drug: Pre-urodynamic Levofloxacin — Levofloxacin 500 mg single dosage 1 hour before the urodynamic examination
  Arms: Pre-urodynamic Levofloxacin
Drug: Post-urodynamic Levofloxacin — Administering once daily Levofloxacin 500 mg for 3 days after urodynamic study
  Arms: Post-urodynamic Levofloxacin

SUMMARY:
This study aims to compare the effectiveness of preoperative single dose of levofloxacin with postoperative levofloxacin for three days on the incidence of urinary tract infections (UTI) after urodynamic examination.

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of preoperative single dose of levofloxacin with postoperative levofloxacin for three days on the incidence of urinary tract infections (UTI) after urodynamic examination. This study uses a randomized single-blind trial design to compare the proportion of posturodynamic UTI in the group receiving preurodynamic single-dose levofloxacin with the group receiving three days - once daily of Levofloxacin posturodynamic. The target population is patients who undergo urodynamic examination at the RSUPN dr. Cipto Mangunkusumo, Siloam ASRI Hospital, and Persahabatan Hospital during the given time.

of the study. The total sample size in this study was determined based on a two-proportion analytical sample calculation formula with type 1 error of 5% and type 2 error of 80%. On the fourth posturodynamic day, urinalysis and urine culture were performed to determine the diagnosis of UTI. To analyze the association between UTI and the treatment group, the chi-square test was used. Results were considered statistically significant if p < 0.05.

The expected results are data on the comparison of the incidence of UTI after urodynamic examination in the group given a single dose of levofloxacin and levofloxacin for three days post-examination.

The incidence of UTI in the group receiving a single preurodynamic dose of levofloxacin compared to the group receiving levofloxacin for three days posturodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Male/female patients > 18 years who have indications for urodynamics
* Willing to participate in research

Exclusion Criteria:

* Allergy to levofloxacin
* History of taking antibiotics in 1 month • Pregnant
* Uncontrolled DM
* Use a urinary catheter
* Having a UTI before urodynamics, based on clinical symptoms and urine examination results
* Refuse to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harrina Erlianti Rahardjo, Professor, Principal Investigator — Indonesia University
Locations (1):
- RS Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
These are the study protocol used in this study
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date
Access Criteria: Anyone who wishes to access the data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The data was collected using a consecutive sampling method until the required number of subjects is reached. The data source of this research is primary data taken from patients who have indications for urodynamic examination at dr. Cipto Mangunkusumo Hospital, Siloam Asri Hospital, and Persahabatan Hospital, Jakarta starting from February 4, 2022
Pre-assignment Details: The inclusion criteria were any above 18-year-old who underwent UDS & were willing to participate in this study. Patients who had at least one of these exclusion criteria were excluded: allergy to levofloxacin, history of antibiotics consumption in 1 month prior to the study, pregnancy, uncontrolled and untreated diabetes mellitus, use of urinary catheter, UTI proved through urinalysis prior to the study, and refusal to participate.
Period: Overall Study
Arm/Group | Pre-urodynamic Levofloxacin | Post-urodynamic Levofloxacin
Started | 67 | 67
Completed | 63 | 63
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-urodynamic Levofloxacin | Post-urodynamic Levofloxacin | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (16) | 53 (17) | 52.5 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 33 | 38 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 63 | 63 | 126
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Urinary Tract Infection
Description: Urinary tract infection is defined based on the result of urinalysis in which one of the following condition present : leukocyes > 5 / high power field, bacteria positive, nitrite positive, and/or positive leukocyte esterase
Time Frame: 4 days after urodynamic
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-urodynamic Levofloxacin | Post-urodynamic Levofloxacin
Number analyzed (Participants) | 63 | 63
Participants | 12 | 13

ADVERSE EVENTS:
Time Frame: After four days of Levofloxacin administration, patients were being assessed for their clinical conditions, such as symptoms related to UTIs, and also adverse events related to Levofloxacin administration and UDS
Description: The adverse events were collected through direct interviews with the patients four days after the procedure. However, one patient reported to the the investigator two days after the procedure due to hematuria.
Arm/Group | Pre-urodynamic Levofloxacin | Post-urodynamic Levofloxacin
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 1/67 | 1/67
Other Adverse Events (participants affected / at risk) | 5/67 | 5/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-urodynamic Levofloxacin (N=67) | Post-urodynamic Levofloxacin (N=67)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) — Patient experienced hematuria two days after urodynamic study
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-urodynamic Levofloxacin (N=67) | Post-urodynamic Levofloxacin (N=67)
Nauseous (Gastrointestinal disorders) | 5 (5) | 5 (5) — Five patients reported that they experience nausea after consuming the antibiotics prescribed

LIMITATIONS AND CAVEATS:
The limitation of the study is that many of the patients with UTIs refuse to undergo urine culture tests due to several reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT05219877/Prot_SAP_000.pdf